CLINICAL TRIAL: NCT07165236
Title: Association of Perioperative Cognitive Dysfunction With Circulating Biomarkers of Neurological Damage in Patients Underging Transurethral Resection of Bladder Tumor
Brief Title: Association of POCD With Circulating Biomarkers in Patients Undergoing TUR of Bladder Tumor
Status: Recruiting | Type: Observational
Sponsor: Osijek University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: POCD
Record Dates: First submitted 2025-03-16; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Cognitive Decline; Urinary Bladder Cancer; Frail; Biomarker; General Anesthesia; Hand Grip Strength; Cognitive Testing; Comorbidities; Demographic Data; Socio-economic Status; Perioperative Complications
Keywords: general anesthesia; postoperative cognitive complications; urinary bladder neoplasm; perioperative period; frail older adult; S100b
MeSH Terms: conditions — Cognitive Dysfunction; Urinary Bladder Neoplasms; Postoperative Cognitive Complications

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adult patients (>18 years) who must undergo transurethral resection of the bladder.: Program operated patients of both sexes would be included. Patients under the age of 18, patients who are unaware, those who cannot give consent for the research, and those who cannot understand the study protocol will be excluded from the study. Patients with proven hypersensitivity to some of the drugs used in the study will also be excluded. Emergency patients, people in a state of shock, septic or severely hemorrhaging patients, and people with previously known neurodevelopmental deficits will not be included in the study.

SUMMARY:
Bladder tumor is one of the most widespread tumors in the world, with increasing prevalence at the global level. One of the procedures in patients with bladder tumors is transurethral resection of the bladder (TURM) most often performed endoscopically under general anesthesia. This patient population has certain characteristics in common. One of them is exposure to common risk factors for the formation of bladder tumors, such as aniline dyes and solvents. These substances are associated with the onset of neurodegeneration and oxidative stress. Smoking is another factor that affects the formation of bladder tumor. A significant part of patients with bladder tumor are an elderly population, which is repeatedly exposed to surgical procedures, with numerous comorbidities, with a high risk of postoperative complications and the development of perioperative cognitive deficits, which can further complicate the postoperative course and further treatment. In the group of patients with a bladder tumor who will undergo TURM, no evaluation of risk factors related to perioperative cognitive deficit was performed, nor was there an examination of the perioperative cognitive deficit itself. In them, the identification of factors for postoperative cognitive disorder is essential. The concept of clinical frailty is becoming more important and relevant when providing healthcare services to patients. The use of the clinical frailty scale as a tool in clinical practice provides information on the adequate direction of care for patients. Decrease in muscle strength can lead to limitations in the functioning of a certain individuals. In recent years muscle strength has come to be a very important component of health, regardless of a person's age and clinical condition.The hand grip test is a test used to measure the maximum isometric strength of the hand and forearm muscles. The MMSE test and MoCA are the most frequently used methods in the detection of cognitive impairment in clinical and research fields. In addition to laboratory indicators of organic function, circulating indicators of neuroinflammation, like S100B and neuron-specific enolase, will be correlated with the patient's cognitive status.So far, no research has been conducted on the dynamics of indicators of organic function, circulating indicators of neuroinflammation, perioperative cognitive changes and clinical fraility in patients undergoing bladder tumor operation.

DETAILED DESCRIPTION:
Bladder tumor is one of the most widespread tumors in the world, with increasing prevalence at the global level. It is the most common malignant disease of the urinary system. One of the procedures in patients with bladder tumors is transurethral resection of the bladder. This procedure is most often performed endoscopically under general anesthesia. The number of patients undergoing this type of procedure is increasing.

This patient population has certain characteristics in common. One of them is exposure to common risk factors for the formation of bladder tumors, such as aniline dyes and solvents. These substances are also associated with the onset of neurodegeneration and oxidative stress. For this reason, cognitive dysfunction can be expected in this patient population in addition to bladder cancer.

Another factor that affects the formation of bladder tumors is smoking. The connection between smoking and the formation of bladder tumors is the presence of carcinogenic substances in the urine of people who smoke, including aromatic amines. Likewise, cigarette smoke itself is harmful, as it also contains numerous carcinogenic substances, which are absorbed from the lungs into the bloodstream, and then reach the bladder via the kidneys. Given that urine is present in the bladder for a long time, its mucosa is exposed to these carcinogenic substances. Carcinogenic substances produced during smoking also lead to an indirect increase in risk, because they damage the immune system of people and lead to the development of inflammatory processes. Smoking is also one of the risk factors associated with the weakening of a person's cognitive status.

A significant part of patients with bladder tumor are an elderly population, which is repeatedly exposed to surgical procedures, with numerous comorbidities, with a high risk of postoperative complications and the development of perioperative cognitive deficits, which can further complicate the postoperative course and further treatment. Postoperative cognitive deficit includes cognitive disorders in the postoperative period, which are associated with numerous complications, which can lead to loss of independence in patients, increased morbidity and mortality, and increase the costs of treatment. In the group of patients with a bladder tumor who will undergo transurethral resection of the bladder, no evaluation of risk factors related to perioperative cognitive deficit was performed, nor was there an examination of the perioperative cognitive deficit itself.

Considering that this is an elderly population, it is expected that some patients will already be frail before the operation with the presence of a significant degree of dementia. In them, the identification of factors for postoperative cognitive disorder is essential, with the aim of taking measures to prevent the deterioration of their impaired general health condition. The concept of clinical frailty is becoming more and more important and relevant when providing healthcare services and healthcare to patients.

Clinical frailty was introduced almost three decades ago as a term in the medical literature, a benchmark for assessing the complex health condition of the elderly and patients with numerous comorbidities. The use of the clinical frailty scale as a tool in clinical practice provides information on the adequate direction of care for patients and information on the further development of health care and health policy. The scale can also help health care providers provide information to patients' families and patients themselves about the risks and benefits of procedures related to the treatment of patients.

Recognition of risk factors and their evaluation are a significant part of perioperative care for patients undergoing surgery under general anesthesia. Risk identification can lead to targeted and directed medical procedures that can be intervened in a timely manner, and reduce the unfavorable clinical outcomes observed after surgical treatment of bladder tumors. Some of these interventions are the recognition and treatment of inflammation, the recognition and correction of anemia, the recognition of clinical frailty, and the implementation of prehabilitation measures in patients undergoing bladder surgery under general anesthesia. Along with them, physical therapy measures could be useful in patients with recognized signs of clinical frailty.

A decrease in muscle strength can lead to limitations in the functioning of a certain individuals. In recent years muscle strength has come to be a very important component of health, regardless of a person's age and clinical condition.

The hand grip test is a test used to measure the maximum isometric strength of the hand and forearm muscles. The test is important for assessing overall upper body strength. Research has shown that hand grip strength is related to important health indicators that include mobility, the overall strength of the person undergoing the hand grip test, the person's cognitive functions, the bone density of the person being tested, but hand grip strength is also related to possible disorders of the cardiovascular system. Improving hand grip strength using strength exercises can help maintain functional independence, especially in older and frail adults. The hand grip test itself is very simple, and in addition, it is also an inexpensive way to assess the overall strength of the upper body, and therefore to detect possible health problems. Monitoring the strength of the hand grip over time can provide valuable insight into the physical abilities of the examined person, and warn of possible disorders that may arise.

In addition to the previously mentioned clinical indicators, laboratory indicators play a significant role in the evaluation of the preoperative condition of the patient and the monitoring of postoperative dynamics. Organ function is regularly assessed in patients by measuring indicators specific to kidney or liver function, such as urea, creatinine, coagulation status, albumin or transaminases.

These indicators could be correlated with clinical frailty and cognitive status. The mini mental state examination test (MMSE) and the cognitive assessment test MoCa (Montreal Cognitive assessment) are the most frequently used methods in the detection of cognitive impairment in clinical and research fields. They are intended as an aid in the clinical examination of the cognitive part of the mental state and are used as instruments for screening for cognitive impairment and monitoring the patient's condition over time. The MMSE is a mental state assessment test, intended as an aid in the clinical evaluation of the cognitive part of the mental state. This test is one of the most commonly used short instruments for screening for cognitive impairment and monitoring the patient's condition over time. The highest number of points on the test is thirty, if a person has less than twenty-four points it is defined as suspected dementia. The MoCa test was originally developed to detect mild cognitive impairment, but it is also used as a screening test for dementia. The total possible test score is thirty points, and a score of twenty-six points or more is considered normal. The MoCA encompasses several different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional abilities, conceptual thinking, calculation and orientation. The time of application of the MoCA test itself is approximately 10 minutes.

In addition to laboratory indicators of organic function, circulating indicators of neuroinflammation, like S100B and neuron-specific enolase, will be correlated with the patient's cognitive status.

So far, no research has been conducted on the dynamics of indicators of organic function, circulating indicators of neuroinflammation, perioperative cognitive changes and clinical fraility in patients undergoing bladder tumor operations under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* adult patients from 18-80 years,
* elective operations of tumor bladder cancer (TUR),
* patients can communicate,
* patients who can sign the information consent and questionnaires

Exclusion Criteria:

* patients under the age of 18,
* patients above 80 years,
* patients who are unable to communicate
* patients who do not understand informed consent for the research,
* patients who are unable to write
* emergency surgery,
* patients with proven hypersensitivity to some of the drugs used in the study
* patients in a state of shock, septic, or hemorrhagic patients with neurodevelopmental disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients, older than 18 years, of both sex, patients that have tumor bladder cancer.
Sampling Method: Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2024-11-28 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
to examine whether the current cognitive state as measured by the Mini-Mental State Examination (MMSE) changes after the patient is exposed to surgery and general anesthesia. | from baseline - 24 hours after surgery- 48 hours after surgery
  Scores are generally interpreted as follows: 25-30: Normal result; 20-25: Mild cognitive impairment; 10-20: Moderate cognitive impairment; 0-10: Severe cognitive impairment. Cognitive test MMSE would be done after before surgery, 24 hours after surgery and 48 hours after surgery
To examine whether the current cognitive state, as measured using the Montreal Cognitive Assessment (MoCA), changes after the patient is exposed to surgery and general anesthesia. | from baseline - 24 hours after surgery- 48 hours after surgery
  The total possible score is 30 points; a score of 26 or above is considered normal. Cognitive test would be done before surgery, 24 hours after surgery, 48 hours after surgery.

SECONDARY OUTCOMES:
to examine changes in s100b in the perioperative period | baseline - 2hours after surgery - 24hours after surgery
  examine chages in s100b preoperatively, 2 hours after surgery, 24 hours after surgery
to examine changes in NSE in the perioperative period | baseline - 2hours after surgery- 24hours after surgery
  examine changes in NSE preoperatively, 2hours after surgery, 24 hours after surgery
to examine changes in IL4 in the perioperative period | baseline - 2hours after surgery- 24hours after surgery
  examine changes in IL4 preoperatively, 2hours after surgery, 24 hours after surgery
to examine changes in iIL6 in the perioperative period | baseline - 2hours after surgery- 24hours after surgery
  examine changes in IL 6 preoperatively, 2hours after surgery, 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Slavica Kvolik, MD, PhD, Study Chair — KBC Osijek
Locations (1):
- Osijek UH, Osijek, Croatia, Croatia

IPD SHARING:
Plan to Share IPD: Yes
data will be available from the author upon request
Supporting Information: Study Protocol
Time Frame: after study complete
Access Criteria: within few days

REFERENCES:
- [Background] Isgro MA, Bottoni P, Scatena R. Neuron-Specific Enolase as a Biomarker: Biochemical and Clinical Aspects. Adv Exp Med Biol. 2015;867:125-43. doi: 10.1007/978-94-017-7215-0_9. PMID 26530364
- [Background] Arevalo-Rodriguez I, Smailagic N, Roque-Figuls M, Ciapponi A, Sanchez-Perez E, Giannakou A, Pedraza OL, Bonfill Cosp X, Cullum S. Mini-Mental State Examination (MMSE) for the early detection of dementia in people with mild cognitive impairment (MCI). Cochrane Database Syst Rev. 2021 Jul 27;7(7):CD010783. doi: 10.1002/14651858.CD010783.pub3. PMID 34313331
- [Background] Picca A, Coelho-Junior HJ, Calvani R, Marzetti E, Vetrano DL. Biomarkers shared by frailty and sarcopenia in older adults: A systematic review and meta-analysis. Ageing Res Rev. 2022 Jan;73:101530. doi: 10.1016/j.arr.2021.101530. Epub 2021 Nov 25. PMID 34839041
- [Background] Carreon T, Hein MJ, Viet SM, Hanley KW, Ruder AM, Ward EM. Increased bladder cancer risk among workers exposed to o-toluidine and aniline: a reanalysis. Occup Environ Med. 2010 May;67(5):348-50. doi: 10.1136/oem.2009.051136. Epub 2009 Nov 2. PMID 19884651
- [Background] Cui HW, Turney BW, Griffiths J. The Preoperative Assessment and Optimization of Patients Undergoing Major Urological Surgery. Curr Urol Rep. 2017 Jul;18(7):54. doi: 10.1007/s11934-017-0701-z. PMID 28589402
- [Background] Demir DO, Doluoglu OG, Yildiz AK, Kacan T, Yazar VM, Demirbas A, Ozgur BC. Effect of Re-TUR time on recurrence and progression in high-risk non-muscle-invasive bladder cancer. Cir Cir. 2022;90(S2):6-12. doi: 10.24875/CIRU.21000905. PMID 36480752
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338